CLINICAL TRIAL: NCT02610426
Title: Exploratory Next Generation Sequencing to Identify Causative Variants for Therapy-Induced Congestive Heart Failure From Breast Cancer Study E5103 Germline DNA Samples
Brief Title: Whole Exome Sequencing in Finding Causative Variants in Germline DNA Samples From Patients With Congestive Heart Failure Receiving Therapy for Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2013-02291; NCI-2013-02291 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E5103T3; E5103T3 (Other: Eastern Cooperative Oncology Group); E5103T3 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2015-11-19; First posted 2015-11-20 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood

GROUPS / COHORTS (1):
- Ancillary-Correlative (whole exome sequencing): Previously collected germline DNA samples are analyzed via whole exome sequencing.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies whole exome sequencing in finding causative variants in germline deoxyribonucleic acid (DNA) samples from patients with congestive heart failure receiving therapy for breast cancer. Studying samples of germline DNA in the laboratory from patients with congestive heart failure receiving therapy for breast cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to congestive heart failure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify, using next generation sequencing, rare variants of large effect size that impact the risk of congestive heart failure (CHF) in patients from the clinical trial ECOG-5103 (E5103).

OUTLINE:

Previously collected germline DNA samples are analyzed via whole exome sequencing.

ELIGIBILITY:
Inclusion Criteria:

* European American patients with DNA available
* European American patients who developed CHF and patients who did not develop CHF following a full course of treatment with an anthracycline and bevacizumab
* African American cases (based on a drop in left ventricular ejection fraction [LVEF] < 50 or a drop from baseline > 20 points) and African American controls

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with breast cancer enrolled on E5103 with or without congestive heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2014-03-25 (Actual); Primary Completion 2100-01-01 (Estimated); Study Completion 2100-01-01 (Estimated)

PRIMARY OUTCOMES:
Identification of rare coding variants of large effect that predict the risk of CHF | Baseline
  Assessed by burden analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan P Schneider, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States